CLINICAL TRIAL: NCT03044548
Title: Improving the Quality of Care for Children With Acute Malnutrition: Cluster Randomised Controlled Trial in West Nile Region, Uganda
Brief Title: Improving the Quality of Care for Children With Acute Malnutrition in Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WHO Collaborating Centre for Maternal and Child Health, Trieste (Other)
Collaborators: CUAMM Doctors for Africa (Unknown)
Responsible Party: Principal Investigator, Marzia Lazzerini, PhD, WHO Collaborating Centre for Maternal and Child Health, Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot 521/2016
Record Dates: First submitted 2016-12-20; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Supportive supervision
  Interventions: Other: Supportive supervision
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Supportive supervision — " Supportive supervision". The specific characteristics of the supportive supervision as intended in this project are outlined below.
  Frequency: Biweekly in the first 3-5 months, than monthly. Duration: approximately 2 hours in each HC at each visit. Provider: local staff (nutritionist, DHO) trained in integrated management acute malnutrition (IMAM) guidelines and in methods of " supportive supervision".
  Receivers: nurses working at HC level with children with malnutrition.
  Reference guidelines:
  • Current National IMAM guidelines
  Attitude and philosophy:
  • Participatory peer-to-peer model based on the Plan - Do- Study- Act quality improvement (QI) Cycle .
  Arms: Experimental

SUMMARY:
This is a cluster RCT in 6 health centres in Uganda, testing supportive supervision to improve health outcomes and quality of care of children with malnutrition

DETAILED DESCRIPTION:
Introduction Malnutrition in children is highly prevalent in West Nile Region. According to a recent analysis of data available from the health management information system (HMIS) and official registers, the health outcomes of children suffering from malnutrition and treated at health center (HC) level in Arua Region are not reaching the international standards (75% cured rate as for the international SPHERE standards). This despite the availability of clear national guidelines for treatment, thus suggesting possible deficiencies in the quality of care provided. Lack of supportive supervision may be one of the reason explaining substandard outcomes.

Methods This is a cluster randomised controlled trail (RCT) with health centers (HC) as unit of randomisation. The six largest HC in Arua district will be randomised in two groups, intervention (quality improvement group) and control. The intervention will aim at improving the quality of care provided at HC level, and as a consequence, the health outcomes of children. The main intervention will consist of enhances nutritional supervision (high frequency supervision, specific to nutritional services), while the control will be standard care (no intervention). Complementary intervention will include training and networking activities for HC staff. Outcomes of the study will include: health outcomes (recovered, non recovered, defaulters, transferred, died); process outcomes (satisfaction and knowledge of staff); cost outcomes (cost for the health system and for the families) and equity outcomes (access to care and health outcomes by wealth quintile).

Relevance of the study The study will inform, with a robust design, about the efficacy and cost-efficacy of a quality improvement intervention for ameliorating the health of children suffering from malnutrition in Uganda.

Currently no other study with RCT design explored the efficacy of supportive supervision as a quality improvement intervention. This study will therefore fill an important knowledge gap.

ELIGIBILITY:
For the primary outcomes, the study sample will consists of children with malnutrition treated at in health center (HC) in Arua district

Inclusion Criteria:

1. Children 6 months-5 years
2. Diagnosis of SAM or MAM according to National criteria (10) SAM: weight-for-height <- 3 standard deviation (SD) from the mean based on the WHO 2006 standards (11).

MAM: weight-for-height <- 2 and > -3 standard deviation (SD) from the mean based on the WHO 2006 growth reference standards .

Exclusion Criteria:

1. Not matching the above criteria for SAM and MAM
2. Refusal to participate/ consent
3. Unable to adhere to study follow up procedures

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 12- 16 weeks
  Rate of cured among children diagnosed with acute malnutrition (SAM and MAM) Cured/discharged is defined as Weight-for-height > -2 standard deviation (SD) from the mean based on the World Health Organisation (WHO) 2006 standards (11) on 2 consecutive visits and no oedema.

SECONDARY OUTCOMES:
Dead rate | 12- 16 weeks
  cases explicitly state as " dead" while in the program
Rate of Not cured | 12- 16 weeks
  Has not reached Cured/discharged criteria in 3 months (4 months for HIV +)
Rate of transferred to ITC (inpatient treatment center) | 12- 16 weeks
  Patients transferred to another outpatient service
Rate of transferred to OTC (outpatient treatment center) | 12- 16 weeks
  Patients transferred to another outpatient service
Rate of defaulted | 12- 16 weeks
  Absent (Not reported or followed up in the community) for 2 consecutive visits.
Quality of data | study start, than every month up to 15 months
  This will be measured by cross-checking data collected from the study data collectors, and data as reported by the staff of the HC
Equity outcomes | study start, than every month up to 15 months
  access to care (supposing that the total population in the coverage area will not change in the intervention period, this will be measured by the crude number of children accessing the HC; efforts will also be made to retrieve, if available, accurate data on changes in the population in the coverage area
Cost | study start, than every month up to 15 months
  Data on cost from the patients (cost of travels to HC, cost of drugs, lab exams etc) and cost for the health services (number of visits in the HC, hospitalisations, foods and other treatments delivered).
Staff satisfaction score | study start, month 6 and month 15
  This will be measured in all staff working with children with malnutrition in the HC participating in the study, using a score system pre-validated for use in Uganda (Hagopian et al, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, PhD, Principal Investigator — WHO CC
Locations (1):
- Arua district, Arua, Uganda

IPD SHARING:
Plan to Share IPD: No